CLINICAL TRIAL: NCT00935025
Title: A Single-center, Single-blind, Randomized, Placebo-controlled, Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics After Single and Multiple Ascending Oral Doses of AZD1305 Extended-release Capsules in Healthy Male Japanese and Caucasian Subjects
Brief Title: AZD1305 Single and Multiple Ascending Dose Study in Healthy Japanese and Caucasian Subjects
Acronym: JMAD
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: D3190C00015
Record Dates: First submitted 2009-07-02; First posted 2009-07-08 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Healthy
Keywords: Phase I; Japanese healthy volunteer; AZD1305; Japanese and Caucasian
MeSH Terms: interventions — tert-butyl (2-(7-(2-(4-cyano-2-fluorophenoxy)ethyl)-9-oxa-3,7-diazabicyclo(3.3.1)non3-yl)ethyl)carbamate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, AZD1305 (Experimental)
  Interventions: Drug: AZD1305
- 2, Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1305 — single and multiple oral doses, extended-release capsule
  Arms: 1, AZD1305
Drug: Placebo — single and multiple oral doses, capsule
  Arms: 2, Placebo

SUMMARY:
This is a phase I, single-blind, randomized, placebo-controlled single and repeated ascending dose study to assess the safety, tolerability and pharmacokinetics with oral doses of AZD1305 extended-release capsules in healthy male Japanese and Caucasian subjects. Three (or four if needed) dose levels will be given to Japanese subjects and one of the doses will also be given to Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese and Caucasian male subjects 20 to 45 years of age inclusive
* Body weight between 50 and 85 kg, inclusive, with a Body Mass Index (BMI) ≥19 to ≤ 27 kg/m2

Exclusion Criteria:

* Clinically significant illness, surgical procedure or trauma, within two weeks preceding the pre-entry visit until first administration of IP, as judged by the investigator
* History of clinically significant gastrointestinal, mental, cardiac, renal or hepatic disorder, or other significant disease as judged by the investigator
* Habitual smoker (daily use) of tobacco or daily use of nicotine-containing products

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Adverse events, ECG variables, vital signs, physical examination, laboratory variables, body temperature and weight | During the study, from screening period to follow-up, 50 days approximately

SECONDARY OUTCOMES:
Pharmacokinetic variables of AZD1305 by assessment of drug concentrations in plasma and urine after single and repeated oral doses | From predose until 48 hrs post last dose

CONTACTS AND LOCATIONS:
Overall Officials: Mark Yen, M.D., Principal Investigator — California Clinical Trials
Locations (2):
- United States (2):
  - Research Site, Glendale, California
  - Research Site, Baltimore, Maryland